CLINICAL TRIAL: NCT02364739
Title: A Randomized Controlled Trial to Evaluate Two Educational Interventions for Increasing Fertility Knowledge and Awareness in Oocyte Donors
Brief Title: Evaluate Educational Interventions for Increasing Fertility Knowledge and Awareness
Acronym: QUESE2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundació Privada Eugin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: QUESE2
Record Dates: First submitted 2013-12-03; First posted 2015-02-18 (Estimated); Last update posted 2015-02-18 (Estimated); Status verified 2015-02

CONDITIONS: Fertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Written information (Experimental): Written information
  Interventions: Other: Written information
- Written and oral information (Experimental): Written and oral information
  Interventions: Other: Written and oral information
- No intervention (No Intervention): Control

INTERVENTIONS:
Other: Written information — Brochure
  Arms: Written information
Other: Written and oral information — Written information consists in a brochure with information about fertility, while oral information consists in a tailored oral explanation about the wrong answers to the pre-test (that is related to the brochure).
  Arms: Written and oral information

SUMMARY:
Fertility knowledge and awareness is considered insufficient in women of reproductive age from developed countries. The objective of this study is to evaluate if educational interventions in oocyte donors increase on their level of fertility knowledge and awareness.

DETAILED DESCRIPTION:
Fertility knowledge and awareness is considered insufficient in women of reproductive age from developed countries. The objective of this study is to evaluate if educational interventions in oocyte donors increase on their level of fertility knowledge and awareness through a RCT. The investigators will evaluate the effect of the interventions through a questionnaire filled in at first visit (pre-test) and at the end of the treatment (post-test); the investigators will compare the increase in the total score between groups.

ELIGIBILITY:
Inclusion Criteria:

* Women candidate to oocyte donation

Exclusion Criteria:

* Previous donations cycles at the center

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 201 (Actual)
Dates: Start 2014-01; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Fertility knowledge increase measured as the difference on total score of the questionnaire at post-test | up to 8 months
  Difference on total score of the questionnaire about fertility knowledge at post-test, that is filled in between 1 and 8 months after the pre-test (i.e. at the end of the donation cycle).

SECONDARY OUTCOMES:
Advancement in the reported ideal age for childbearing at post-test | up to 8 months
  Difference on the reported ideal age for childbearing at post-test, respect to the pre-test

CONTACTS AND LOCATIONS:
Overall Officials: Désirée García, Principal Investigator — Fundació Privada Eugin
Locations (1):
- Clinica EUGIN, Barcelona, Barcelona, Spain